CLINICAL TRIAL: NCT05701553
Title: Phase I/II Study of Anti-PD-1/PD-L1 Antibodies Combined With S-adenosyl-methionine in Patients With Advanced-Stage Hepatocellular Carcinoma
Brief Title: Anti-PD-1/PD-L1 Antibodies Plus S-adenosyl-methionine Treatment in Patients With Advanced-Stage Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2022-118
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Anti-PD-1 antibody; Anti-PD-L1 antibody; SAM
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — S-Adenosylmethionine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood specimen and tissue samples will be collected performing related experiments including metabolomics analysis, lipidomics analysis and flow cytometry etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-PD-1/PD-L1 antibodies and S-adenosyl-methionine combination: Drug: Anti-PD-1/PD-L1 Intravenous injection for at least 6 months
  Drug: S-adenosyl-methionine Taken orally for at least 6 months
  Interventions: Drug: Anti-PD-1/PD-L1; Drug: S-Adenosyl-Methionine

INTERVENTIONS:
Drug: Anti-PD-1/PD-L1 — Intravenous injection at indicated dose for at least 6 months
Drug: S-Adenosyl-Methionine — Taken orally at indicated dose for at least 6 months
  Other Names: SAM

SUMMARY:
This study is being done to analyze the safety, tolerability, and efficacy of treatment using combination of SAM and anti-PD-1/PDL1 antibodies for patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a study of combination anti-PD-1/PD-L1 antibodies and S-adenosyl-methionine (SAM) for adult patients (≥18) with advanced hepatocellular carcinoma.

SAM is a compound found naturally in the body and is available as a dietary supplement in the U.S. SAM is a prescription drug in China treating liver disease and advanced HCC with poor liver function under certain circumstances. Also, SAM has recently been shown to play a key role regulating cancer cell proliferation trough epigenetic pathway.

Anti-PD-1/PD-L1 antibodies (including pembrolizumab, nivolumab, sintilimab, toripalimab, camrelizumab, tislelizumab and atezolizumab etc.) are given intravenously at assigned dose. Treatment may continue until disease progression, intolerable toxicity, or consent withdrawal.

This study is aimed to evaluate the safety and efficacy of the combination of SAM and PD-1/PD-L1 monoclonal antibody in unresectable late-stage HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male or female
2. Advanced hepatocellular carcinoma (cannot be removed or metastasized) diagnosed clinically or pathologically, at least one measurable lesion without local treatment, Child-Pugh A ;Barcelona Clinic Liver Cancer(BCLC) staging is stage B or C
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
4. Patient has given written informed consent.
5. The function of important organs meets the requirements
6. Expected survival ≥12 weeks
7. Non-surgical sterilization or women of childbearing age need to use a medically-accepted contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid Hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included);
2. The patient is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg / day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment;
3. Have clinical symptoms or disease that are not well controlled;
4. Significant clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to randomization;
5. Arterial/venous thrombosis in the first 6 months of randomization
6. According to the investigator, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory abnormalities.#with family or social factors, it will affect the safety of patients.
7. Liver tumor burden greater than 50% of the total liver volume, or patients who have previously undergone liver transplantation;Known for a history of central nervous system metastasis or hepatic encephalopathy;Severe allergic reactions to other monoclonal antibodies;

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Advanced hepatocellular carcinoma (cannot be removed or metastasized) diagnosed clinically or pathologically, at least one measurable lesion without local treatment, Child-Pugh A ;Barcelona Clinic Liver Cancer(BCLC) staging is stage B or C
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last treatment dose
  Safety will be monitored by addressing and recording all adverse events (AEs), serious adverse events (SAEs) and specific laboratory abnormalities (worst grade). Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

SECONDARY OUTCOMES:
Objective response rate(ORR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Progression free survival(PFS) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
To the relief time (TOR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Duration of relief(DOR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Disease Control Rate (DCR) | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
6-month survival rate | 6 months
  Evaluated by researchers based on the RECIST 1.1 standard
12-month survival rate | 12 months
  Evaluated by researchers based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou J, Sun H, Wang Z, Cong W, Wang J, Zeng M, Zhou W, Bie P, Liu L, Wen T, Han G, Wang M, Liu R, Lu L, Ren Z, Chen M, Zeng Z, Liang P, Liang C, Chen M, Yan F, Wang W, Ji Y, Yun J, Cai D, Chen Y, Cheng W, Cheng S, Dai C, Guo W, Hua B, Huang X, Jia W, Li Y, Li Y, Liang J, Liu T, Lv G, Mao Y, Peng T, Ren W, Shi H, Shi G, Tao K, Wang W, Wang X, Wang Z, Xiang B, Xing B, Xu J, Yang J, Yang J, Yang Y, Yang Y, Ye S, Yin Z, Zhang B, Zhang B, Zhang L, Zhang S, Zhang T, Zhao Y, Zheng H, Zhu J, Zhu K, Liu R, Shi Y, Xiao Y, Dai Z, Teng G, Cai J, Wang W, Cai X, Li Q, Shen F, Qin S, Dong J, Fan J. Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2019 Edition). Liver Cancer. 2020 Dec;9(6):682-720. doi: 10.1159/000509424. Epub 2020 Nov 11. PMID 33442540
- [Background] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Background] Lu SC, Mato JM. S-adenosylmethionine in liver health, injury, and cancer. Physiol Rev. 2012 Oct;92(4):1515-42. doi: 10.1152/physrev.00047.2011. PMID 23073625
- [Background] Kraeuchi K, Rudolph K, Wirz-Justice A, Feer H. Similarities in feeding behavior of chronic methamphetamine treated and withdrawn rats to VMH lesioned rats. Pharmacol Biochem Behav. 1985 Dec;23(6):917-20. doi: 10.1016/0091-3057(85)90092-9. PMID 4080776